CLINICAL TRIAL: NCT06253130
Title: A First-in-human, Phase 1/2, Open-label, Multi-center, Dose-escalation, Dose-optimization, and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Anti-tumor Activity of PARP1 Selective Inhibitor, IMP1734, as Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A First-in-human Study of PARP1 Selective Inhibitor, IMP1734, in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Collaborators: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EIK1003-001 (IMP1734-101); 2023-509230-19 (EudraCT Number)
Record Dates: First submitted 2024-01-27; First posted 2024-02-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
Keywords: EIK1003; EIK1003-001; IMP1734

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): IMP1734 monotherapy; oral tablet(s) daily (except for the single-dose period). The maximum trial duration is 3 years after the last participant's first treatment in the trial.
  Interventions: Drug: IMP1734

INTERVENTIONS:
Drug: IMP1734 — PARP1 selective inhibitor

SUMMARY:
This study will evaluate the preliminary efficacy of IMP1734 in patients with recurrent advanced/metastatic breast cancer, ovarian cancer and metastatic castrate resistant prostate cancer (mCRPC) with deleterious/suspected deleterious mutations of select homologous recombination repair (HRR) genes.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability and preliminary efficacy of IMP1734 as monotherapy in patients with recurrent, advanced/metastatic solid tumors. The study consists of 3 parts: Dose escalation, Dose Optimization and Dose expansion.

In dose escalation (Part1), the study will identify the maximum tolerated dose (MTD) or maximum achievable dose (MAD) in solid tumor.

In dose optimization (Part 2), the study will further evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and anti-tumor activity of select doses of IMP1734.

In dose expansion (Part 3) the recommended dose escalation (RDE) of IMP1734 monotherapy will be evaluated in patients with recurrent, advanced/metastatic breast cancer, ovarian cancer and mCRPC with deleterious/suspected deleterious mutations of select homologous recombination repair (HRR) gene mutations.

ELIGIBILITY:
Key Inclusion Criteria

* Breast cancer; must have received at least one prior chemotherapy in neoadjuvant/adjuvant/metastatic setting, must have received hormonal therapy if HR+,
* HGSOC or high grade endometrioid EOC, fallopian tube or primary peritoneal cancer; must have received at least one prior platinum-based chemotherapy for advanced disease
* mCRPC with ongoing ADT, must have received NHA and up to 1 prior line of taxane chemotherapy
* Age ≥ 18 years at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate organ function
* Life expectancy ≥ 12 weeks
* Should have evaluable disease as defined by RECIST1.1 and/or CA125 or PSA
* Female subjects of childbearing potential and male subjects must agree to use an effective method of contraception from study entry up to 6 months after the last dose of IMP1734
* deleterious or suspected deleterious germline or somatic mutations of select HRR genes
* up to 1 prior line of PARP inhibitor containing treatment

Key Exclusion Criteria:

* Any investigational or approved anti-cancer therapies administered within 28 days/ before the first dose of IMP1734
* Have received prior PARP1 selective inhibitors
* Mean resting QTcF > 470 ms or QTcF < 340 ms
* Active or untreated central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Infections

  - An active hepatitis B/C infection
* Any known predisposition to bleeding
* Unable to swallow oral medications OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition that might impair the bioavailability

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events, treatment emergent adverse events or serious adverse events | Consent to 30 + 7 days post last dose of IMP1734
  Number of subjects reporting adverse events or serious adverse events which include any abnormal clinical events, laboratory assessments outside of normal clinical range, abnormal vital signs observed, and any abnormal ECG parameters
Maxim Tolerated Dose or Recommended Dose for Expansion | DLT period is from the first dose of the study drug until the last day of the first cycle
  Number of patients that experience a DLT or any toxicity which occurs from the time of the first dose of study drug until the end of cycle 1, which is deemed unrelated to the disease.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of IMP1734 | Through study completion, up to 3 years
  Peak plasma concentration (Cmax)
Pharmacokinetic parameters of IMP1734 | Through study completion, up to 3 years
  Time to peak drug concentration (Tmax)
Pharmacokinetic parameters of IMP1734 | Through study completion, up to 3 years
  Area under the curve (AUC) will be defined
Overall Response Rate | Through study completion, up to 3 years
  Percentage of participants who have CR/PR per RECIST v1.1,and/or CA125 response per GCIG criteria (ovarian cancer), and/or PSA response per PCWG3 criteria

OTHER OUTCOMES:
Characterization of the pharmacodynamic changes due to IMP1734 | Through study completion, up to 3 years
  Evaluation of serial pharmacodynamic changes across multiple doses of IMP1734

CONTACTS AND LOCATIONS:
Overall Officials: Viola Chen, MD, Study Director — Eikon Therapeutics
Locations (54):
- United States (23):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - Hoag Health Center Irvine, Irvine, California
  - University California Irvine, Irvine, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Sarah Cannon Research Institute Health One, Denver, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Advent Health Research Institute, Celebration, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota-Clinical Research Unit, Minneapolis, Minnesota
  - Washington University - Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Cayuga Medical Center, Ithaca, New York
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Medical University of South Carolina (MUSC) - Hollings CC, Charleston, South Carolina
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - Sarah Cannon Research Institue Oncology, Nashville, Tennessee
  - START - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
- Australia (6):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Mater Cancer Care Centre, Mater Misericordiae Limited, South Brisbane, Queensland
  - Gold Coast Private Hospital, Southport, Queensland
  - Macquarie University, Sydney, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peninsula and south eastern haematology and oncology group, Frankston, Victoria
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre-University Health Network, Toronto, Ontario
- China (4):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Chongqing University Cancer Hospital, Chongqing
  - Zhejiang Cancer Hospital, Hangzhou
  - Fudan University Shanghai Cancer Center, Shanghai
- Righospitalet, Copenhagen, Denmark
- France (3):
  - Hospices Civils de Lyon - CHU Lyon Sud, Pierre-Bénite, Rhone
  - CLCC François Baclesse, Caen
  - Institut Gustave Roussy, Villejuif
- South Korea (3):
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Gachon University - Gil Medical Center, Incheon, Namdong-gu
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (10):
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Clínica Universidad de Navarra - Hospital, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Fundacion MD Anderson Cancer Center, Madrid
  - START Madrid Fundación Jiménez Díaz, Madrid
  - START-CIOCC HM Sanchinarro Hospital, Madrid
  - Universidad De Sevilla - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia - INCLIVA, Valencia